CLINICAL TRIAL: NCT04501653
Title: Precision Functional Brain Mapping to Understand the Mechanisms of Psilocybin
Brief Title: Precision Functional Brain Mapping in Psilocybin
Acronym: Psilocybin PFM
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Ginger E Nicol, Professor of Psychiatry, Washington University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 202002165; GF0010787 (Other: Washington University)
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2024-10

CONDITIONS: Psilocybin
MeSH Terms: interventions — Psilocybin; psilocin; Methylphenidate

STUDY DESIGN:
Intervention Model Description: Participants will undergo a baseline imaging session, followed by a blinded drug session with psilocybin 25mg, or methylphenidate (MTP) 40mg. Participants will then have a "between" imaging session without medication, followed by another medication imaging session with the agent not used in the first medication session. This will be followed by a final imaging session without medication.
Who Masked: Participant
Masking Description: Participants will be aware that they are receiving either psilocybin or methylphenidate at each medication imaging session, but will not be told in what order they will receive study medication (psilocybin first versus methylphenidate first).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Psilocybin first (Experimental): Participants will receive 25 mg of psilocybin at the first of two neuroimaging sessions, taken orally in capsule form. Participants in this arm will receive the control drug (methylphenidate) at their second drug exposure neuroimaging session.
  Interventions: Drug: Psilocybin; Drug: Methylphenidate
- Methylphenidate first (Active Comparator): Participants in this group will be randomized to receive 40 mg of methylphenidate at the first of two neuroimaging sessions, taken orally in capsule form. Participants in this arm will receive the active comparator (psilocybin) at their second drug exposure neuroimaging session.
  Interventions: Drug: Psilocybin; Drug: Methylphenidate

INTERVENTIONS:
Drug: Psilocybin — Psilocybin is a naturally occurring psychedelic compound produced by psilocybin mushrooms, and has been shown to have antidepressant and anti-anxiety effects after one dose of 25 mg. Common side effects are slight elevations in blood pressure and heart rate. Participants will be randomized to receive either psilocybin or control at two separate imaging timepoints in this study.
  Other Names: psilocin
Drug: Methylphenidate — Methylphenidate is a stimulant medication used to treat attention deficit hyperactivity disorder (ADHD) and narcolepsy, and is used as an active control for this study because it is metabolized similarly to psilocybin and has similar effects on heart rate and blood pressure. Participants will be randomized to receive either psilocybin or control at two separate imaging timepoints in this study.
  Other Names: Metadate, Methylin, Ritalin, Concerta

SUMMARY:
This project will employ functional brain imaging to study the mechanism and immediate and long-term effects of psilocybin, a serotonin receptor 2A agonist, on cortical and cortico-subcortical brain networks in healthy adults.

DETAILED DESCRIPTION:
Psilocybin shows promise as a safe, transformational therapeutic across several psychiatric conditions. However, little is know about its mechanism of action. This study aims to establish a neuroimaging paradigm for use in future clinical research testing the effectiveness of psilocybin in various clinical applications.

In this study, we will assess both acute (during psilocybin exposure) and sustained (one week post-exposure) effects of 5-HT2A receptor agonism on brain circuits using resting state functional connectivity and precision functional mapping (PFM). Using a randomized, controlled crossover study design, a small number of healthy volunteers will receive either psilocybin or methylphenidate (MTP) and will undergo MRI (structural, task, blood flow, extended resting state). After two weeks, participants will return for a second exposure with the alternate of what they received in the first session. This study involves up to five separate imaging sessions.

Functional connectivity will be measured using the following PFM approach:

1. Extended functional magnetic resonance imaging (fMRI) image acquisition
2. Aggressive data cleaning
3. Analysis designed to examine functional brain connectivity at the individual level

This will allow us to map the effects of 5-HT2A receptor agonism on cortical and cortico-subcortical brain networks at the individual level with precision that is unparalleled in the current literature. This is the first step in developing a precision neuroimaging approach for mechanistic understanding of psilocybin's therapeutic effects.

If successful, this pharmacoimaging paradigm will have potential utility across psychiatric conditions, allowing us to better understand whether and how psilocybin might "bend the curve" in treatment course, preventing persistent suffering, disability, and suicide.

ELIGIBILITY:
Inclusion Criteria:

1. men and woman between 18 and 40 years of age;
2. Have used a psychedelic substance within the previous 5 years but not within the last 6 months
3. No active psychiatric conditions requiring treatment with psychotropic medications (may be included if psychiatric condition is stable and participant is willing to discontinue medication for 1 month prior to participation with permission from their treating provider);
4. Able to provide informed consent.

Exclusion Criteria:

1. Presence of medical conditions that may confound results of imaging study or that are contraindications to psilocybin exposure (e.g. neurological, renal, hypertension, metabolic or cardiovascular disease or pregnancy);
2. No prior exposure to classic psychedelics (psilocybin, LSD, ayahuasca, mescaline);
3. Presence of psychiatric conditions that may confound interpretation of results or that are contraindications to psilocybin exposure (e.g. major mood disorder, current substance use disorder, personal or immediate family history (parents, siblings) of any schizophrenia spectrum disorders);
4. Use of psychotropic medication during the study;
5. Presence of contraindications to MRI scanning (implantable devices, bone hardware, IUD).
6. Prior adverse reactions to psychedelics, based on the Challenging Experiences Questionnaire administered during initial screening

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-03-19 (Actual); Study Completion 2023-03-19 (Actual)

PRIMARY OUTCOMES:
Functional Connectivity | 1 week
  Our overall goal is to use a Functional Connectivity (very long scans to produce individual connectomes) to examine the effects of psilocybin on cortical and cortico- subcortical brain networks that could explain its rapid and sustained behavioral effects.

SECONDARY OUTCOMES:
Mystical Experiences | 1 week
  Measured using Persisting Effects Questionnaire
Personality Change | 1 week
  Measured using International Personality Item Pool-Five-Factor Model

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No